CLINICAL TRIAL: NCT00041847
Title: Gene-Environment Interaction in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 11126-CP-001
Record Dates: First submitted 2002-07-18; First posted 2002-07-22 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: gene; environment; occupation; diet; interaction
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to determine whether certain environmental factors, namely occupational exposures and diet, have a greater effect on prostate cancer risk in the presence of selected inherited genetic factors.

ELIGIBILITY:
men diagnosed with prostate cancer before age 70 and race/age frequency matched healthy controls

Max Age: 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2001-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States